CLINICAL TRIAL: NCT04064853
Title: Childrens' Experiences of Pain in Conjunction With Tooth Extraction - a Grounded Theory
Brief Title: Childrens' Experiences of Pain in Conjunction With Tooth Extraction - a Grounded Theory Study
Status: Completed | Type: Observational
Sponsor: Malmö University (Other)
Responsible Party: Principal Investigator, Henrik Berlin, DDS, senior lecturer, Malmö University
Other Study IDs: GT dental pain Malmo U
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Attitude; Pain, Postoperative; Pain, Procedural; Child; Adolescent; Tooth Extraction
Keywords: grounded theory; child; adolescent; postoperative pain; procedural pain; tooth extraction
MeSH Terms: conditions — Behavior; Pain, Postoperative; Pain, Procedural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a qualitative study, using Grounded Theory. The aim is to deepen our knowledge about how children perceive pain in conjunction with dental treatment; tooth extractions in particular. What increases, and what decreases, the risk of children experiencing pain; and how do they perceive dental treatments where pain might occur, either as procedural pain, or postoperatively?

DETAILED DESCRIPTION:
BACKGROUND: Pain in conjunction with dental treatment should be avoided as much as possible, when treating children. Many dental procedures may result in procedural and/or postoperative pain. There is a well-documented relationship between perceived pain during/after dental treatment, and the development of dental fear and anxiety. This may lead to suffering for the patient and accelerating treatment-costs for society. Despite this, research on children and pain is scarce. Systematic review shows a lack of studies on oral analgesics and their possibility to reduce/prevent pain. There is a need for randomized clinical trials regarding different treatments and effect of analgesics. However, before such research can be undertaken, one important piece is missing; an understanding on how children and adolescents perceive dental treatment and the possible pain afterwards. The aim of this study is to elucidate how children perceive dental treatment and pain after tooth extractions.

METHODS: This is a qualitative study using Grounded Theory (GT). Children aged 10-15 years, who needs teeth extracted prior orthodontic treatment, will be consecutively enrolled if the legal guardians signs the informed consent-form and the child assents to participate. Tooth extractions will then be performed by another dentist than the one doing the interviews with the children. A treatment protocol, in accordance with today standardized practice, for the extractions will be followed. No extra dental treatment is performed, rather this is a part of the whole treatment plan for orthodontic treatment. In-depth interview will be performed with the children 1-2 weeks after tooth extraction, at a place convenient for the child/family. If the participant wishes to, they can be accompanied by their legal guardian during the interview. The questions will focus on their experiences of the tooth extraction, perceived pain, pain management, coping strategies, and previous experiences of pain and how they handled it then. Each interview is calculated to take approximately one hour. In Grounded Theory no sample size calculation is applicable. Participants will be included until saturation in data is reached, i.e. no new information can be obtained. In GT this is often achieved after 10-15 interviews, but when it involves children it is not unlikely that the number of participants will be closer to 20, since there is a risk of the interviews not being so "rich". All interviews will be tape recorded, and without further delay, the interviews will be transcribed. Data analyses and data collection will be done parallel with each other. The transcribed interviews will be analyzed, where codes will be identified. These codes will then merge into different preliminary categories. In the following axial coding process, each category will be further developed by identifying dimensions and characteristics (sub-categories). Relations between data and categories is sought for, and hereby a new whole is created. Selective coding will lead to data saturation and validation. Saturation can also be achieved by already retrieved data being re-coded.

KNOWLEDGE GAINS: GT is a theory generating method. This is especially suitable for research areas where theories are scarce or completely lacking. A lot of research within the medical and dental field today, takes the perspective of the investigator, and far too seldom is those directly affected (i.e. the patient), involved. From an ethical point of view, it is important to include children and adolescents if the research is targeting this group. If knowledge about how children and adolescents perceive pain is gained, this will be an important piece in assembling the puzzle of research strategies related to pain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* In need of extraction of permanent premolars prior orthodontic treatment

Exclusion Criteria:

* If sedation is needed to be able to comply with dental treatment
* Do not understand Swedish language

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 10-15 years of age, identified as eligable according to inclusion and exclusion criteria, during first visit to orthodontist, working in city of Malmö, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Children's experiences during and after tooth extraction, and it's consequences | Fall 2019
  After tooth extraction, on orthodontic indications, participants, 10-15 years of age, are interviewed. The interviews are transcribed and analyzed, identifying codes, which will be clustered into categories. Through different types of methods, used in Grounded Theory, core categories will be identified which together with other categories and sub-categories, will answer the question "what is all this about?".

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Berlin, DDS, Principal Investigator — Malmö University, Faculty of Odontology
Locations (1):
- Faculty of Odontology, Malmö University, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared.

REFERENCES:
- [Background] Berlin H, List T, Ridell K, Davidson T, Toft D, Klingberg G. Postoperative pain profile in 10-15-year-olds after bilateral extraction of maxillary premolars. Eur Arch Paediatr Dent. 2019 Dec;20(6):545-555. doi: 10.1007/s40368-019-00425-9. Epub 2019 Apr 8. PMID 30963511
- [Background] Berlin H, List T, Ridell K, Klingberg G. Dentists' attitudes towards acute pharmacological pain management in children and adolescents. Int J Paediatr Dent. 2018 Mar;28(2):152-160. doi: 10.1111/ipd.12316. Epub 2017 Jul 10. PMID 28691744
- [Background] Charmaz K. Grounded theory. In: Smith JA, Harre R, van Langenhove L, eds. Rethinking methods in psychology, 2nd ed. London: Sage Publications, 1995; 27-49.
- [Background] Charmaz K. Grounded theory. Objectivist and constructivist methods. In: Denzin NK, Lincoln YS, eds. Handbook of qualitative research, 2nd ed. Thousand Oaks, CA: Sage, 2000; 509-535.
- [Background] Dellve L, Henning Abrahamsson K, Trulsson U, Hallberg LR-M. Grounded theory in public health research. In: Hallberg LR-M, ed. Qualitative methods in public health research: theoretical foundations and practical examples. Lund: Studentlitteratur, 2002; 137-173.
- [Background] Glaser B, Strauss A. The discovery of grounded theory: strategies for qualitative research. New York: Aldine de Gruyter, 1967.
- [Background] Ashley PF, Parekh S, Moles DR, Anand P, MacDonald LC. Preoperative analgesics for additional pain relief in children and adolescents having dental treatment. Cochrane Database Syst Rev. 2016 Aug 8;2016(8):CD008392. doi: 10.1002/14651858.CD008392.pub3. PMID 27501304